CLINICAL TRIAL: NCT01341626
Title: Juvenile Justice Girls: Pathways to Adjustment and System Use in Young Adulthood
Brief Title: Juvenile Justice Girls Randomized Control Trial: Young Adult Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); University of Oregon (Other)
Responsible Party: Principal Investigator, Leslie D. Leve, Study Principal Investigator, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA024672 (NIH); R01DA015208 (NIH); R01MH054257-01 (NIH); R03MH091611 (NIH)
Record Dates: First submitted 2011-04-06; First posted 2011-04-26 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Delinquency; Drug Use
Keywords: delinquency; drug use; HIV risk behavior; economic costs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Foster Care Oregon (TFCO) (Experimental): Youth are placed individually in well-trained and supervised foster homes. Basic components include: (a) daily telephone contact with TFCO parents using the Parent Daily Report; (b) weekly foster parent group meetings focused on supervision, training in parenting practices, and support; (c) an individualized behavior management program implemented daily in the home by foster parent; (d) individualized skills training for the youth; (e) family therapy for aftercare family focused on parent management strategies; (f) close monitoring of school attendance, performance, and homework completion; (g) case management to coordinate TFCO, family, peer, and school settings; (h) 24-hour on-call staff availability to TFCO and biological parents; and (i) psychiatric consultation.
  Interventions: Behavioral: Treatment Foster Care (TFCO)
- Group Care (Active Comparator): Group Care is the usual service for youth placed in out-of-home care for chronic delinquency in Oregon. These programs represented typical services for girls being referred to out-of-home care by the juvenile justice system and had 2-51 youth in residence (M = 21) and 1-50 staff members (Mdn = 2); most also had onsite schooling. Although the programs differed somewhat in theoretical orientations, 86% reported that they endorsed a specific treatment model, of which the primary philosophy was a behavioral (70%), eclectic (26%), or family-style therapeutic approach (4%).
  Interventions: Behavioral: Group Care

INTERVENTIONS:
Behavioral: Treatment Foster Care (TFCO) — Youth placed individually in well-trained and supervised foster homes. Basic components: (a) daily telephone contact with TFCO parents; (b) weekly foster parent group meetings focused on supervision, training in parenting practices, and support; (c) an individualized behavior management program implemented daily in the home by foster parent; (d) individualized skills training for the youth; (e) family therapy for aftercare family focused on parent management strategies; (f) close monitoring of school attendance, performance, and homework completion; (g) case management to coordinate TFCO, family, peer, and school settings; (h) 24-hour on-call staff availability to TFCO and biological parents; and (i) psychiatric consultation. Services typically last approximately 6 months.
  Other Names: Multidimensional Treatment Foster Care
  Arms: Treatment Foster Care Oregon (TFCO)
Behavioral: Group Care — Group Care is the usual service for youth placed in out-of-home care for chronic delinquency in Oregon. These programs represented typical services for girls being referred to out-of-home care by the juvenile justice system and had 2-51 youth in residence (M = 21) and 1-50 staff members (Mdn = 2); most also had onsite schooling. Although the programs differed somewhat in theoretical orientations, 86% reported that they endorsed a specific treatment model, of which the primary philosophy was a behavioral (70%), eclectic (26%), or family-style therapeutic approach (4%). Services typically last approximately 6 months.
  Arms: Group Care

SUMMARY:
This study is a young adult follow-up of 166 females who originally participated in an RCT during adolescence due to their involvement in the juvenile justice system.

DETAILED DESCRIPTION:
Females under age 18 years old are the fastest-growing segment of the juvenile justice population and are at risk for negative co-occurring outcomes including drug abuse, HIV/STI risk, criminal behavior, and educational failure. As they enter young adulthood, this constellation of behaviors puts them at heightened risk for early parenthood and subsequent involvement in the child welfare system (for their parenting behaviors) and the adult corrections system (for criminal behaviors). Such system involvement is costly, and its prevention would be of great significance to public health; however, very little is known about factors leading to females' success/failure in young adulthood and factors that might prevent involvement in these two public systems. This study aims to further our understanding of the pathways to and the prevention of HIV/STI risk, drug use, and child welfare and adult corrections involvement by following-up 166 women who participated in two randomized intervention trials aimed at reducing delinquency during adolescence. In the original studies, juvenile justice girls who had been referred for out-of-home placement due to chronic delinquency were randomly assigned to services as usual or to Treatment Foster Care Oregon (TFCO, formerly known as MTFC). Efficacy of the intervention with this sample has been shown at 12- and 24-month follow-ups on criminal referral rates, days spent in locked settings, deviant peer associations, educational engagement, and pregnancy prevention. The investigators propose to examine the developmental pathways for these juvenile justice girls into young adulthood (ages 21-28 years) using innovative data collection and data analytic techniques, with foci on the long-term effects of TFCO, the mediators of young adult adjustment and child welfare/corrections involvement, and the cost effectiveness and cost avoidance of TFCO on these outcomes. The overarching aim is to identify potential targets for subsequent intervention. One in-person assessment is proposed with each female and her current romantic partner (if she has one); in addition, telephone interviews will be conducted every 6 months for the duration of the study, and system data from child welfare and adult corrections will be collected.

ELIGIBILITY:
Inclusion Criteria:

* female
* 13-17 years old
* at least one criminal referral in the prior year
* court-mandated placement in out-of-home care

Exclusion Criteria:

* Currently pregnant

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 1997-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Delinquency | Months 12, 24, 36, and young adulthood (ave. of 7 year follow-up + 10 year follow-up)
  Measured as self-reported criminal activity and count of official arrests and criminal referrals
substance use | Months 12, 24, 36 and young adulthood (ave. of 7-year follow-up + 10 year follow-up)
  Measured via self-reported use and diagnostic interview assessment

SECONDARY OUTCOMES:
HIV risk behavior | Months 12, 24, 36 and young adulthood (ave. of 7-year follow-up)
  Measured as self-reported engagement in sexual behaviors
economic costs | young adulthood (age 18-28; average of 7-year follow-up)
  Measured by comparing the costs of intervention delivery relative to the two intervention programs relative to costs incurred through time in detention, jail, and prison; relative to costs incurred due to child welfare involvement; and relative to symptom counts on self-report inventories.
Depression | Months 6, 12, 18, 24 and Young Adult (average 7 year follow-up)
  Measured on the CESD depression inventory and the Brief Symptom Inventory, and via diagnostic interview

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Leve, PhD, Principal Investigator — University of Oregon
Locations (2):
- United States (2):
  - Oregon Social Learning Center, Eugene, Oregon
  - University of Oregon, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harold GT, Kerr DC, Van Ryzin M, DeGarmo DS, Rhoades KA, Leve LD. Depressive symptom trajectories among girls in the juvenile justice system: 24-month outcomes of an RCT of Multidimensional Treatment Foster Care. Prev Sci. 2013 Oct;14(5):437-46. doi: 10.1007/s11121-012-0317-y. PMID 23417664
- [Result] Van Ryzin MJ, Leve LD. Affiliation with delinquent peers as a mediator of the effects of multidimensional treatment foster care for delinquent girls. J Consult Clin Psychol. 2012 Aug;80(4):588-96. doi: 10.1037/a0027336. Epub 2012 Feb 20. PMID 22352857
- [Result] Kerr DC, Leve LD, Chamberlain P. Pregnancy rates among juvenile justice girls in two randomized controlled trials of multidimensional treatment foster care. J Consult Clin Psychol. 2009 Jun;77(3):588-93. doi: 10.1037/a0015289. PMID 19485598
- [Result] Chamberlain P, Leve LD, Degarmo DS. Multidimensional treatment foster care for girls in the juvenile justice system: 2-year follow-up of a randomized clinical trial. J Consult Clin Psychol. 2007 Feb;75(1):187-93. doi: 10.1037/0022-006X.75.1.187. PMID 17295579
- [Result] Leve LD, Chamberlain P, Reid JB. Intervention outcomes for girls referred from juvenile justice: effects on delinquency. J Consult Clin Psychol. 2005 Dec;73(6):1181-5. doi: 10.1037/0022-006X.73.6.1181. PMID 16392991
- [Result] Level LD, Chamberlain P. Association with delinquent peers: intervention effects for youth in the juvenile justice system. J Abnorm Child Psychol. 2005 Jun;33(3):339-47. doi: 10.1007/s10802-005-3571-7. PMID 15957561
- [Result] Leve LD, Chamberlain P. A Randomized Evaluation of Multidimensional Treatment Foster Care: Effects on School Attendance and Homework Completion in Juvenile Justice Girls. Res Soc Work Pract. 2007 Nov 1;17(6):657-663. doi: 10.1177/1049731506293971. PMID 18159224
- [Result] Rhoades KA, Chamberlain P, Roberts R, Leve LD. MTFC for High Risk Adolescent Girls: A Comparison of Outcomes in England and the United States. J Child Adolesc Subst Abuse. 2013 Nov 1;22(5):435-449. doi: 10.1080/1067828X.2013.788887. PMID 24003300
- [Result] Leve LD, Kerr DC, Harold GT. Young Adult Outcomes Associated with Teen Pregnancy Among High-Risk Girls in an RCT of Multidimensional Treatment Foster Care. J Child Adolesc Subst Abuse. 2013 Sep 1;22(5):421-434. doi: 10.1080/1067828X.2013.788886. PMID 24453470
- [Result] Poulton R, Van Ryzin MJ, Harold GT, Chamberlain P, Fowler D, Cannon M, Arseneault L, Leve LD. Effects of multidimensional treatment foster care on psychotic symptoms in girls. J Am Acad Child Adolesc Psychiatry. 2014 Dec;53(12):1279-87. doi: 10.1016/j.jaac.2014.08.014. Epub 2014 Sep 16. PMID 25457926
- [Result] Kerr DC, DeGarmo DS, Leve LD, Chamberlain P. Juvenile justice girls' depressive symptoms and suicidal ideation 9 years after Multidimensional Treatment Foster Care. J Consult Clin Psychol. 2014 Aug;82(4):684-93. doi: 10.1037/a0036521. Epub 2014 Apr 14. PMID 24731234
- [Result] Rhoades KA, Leve LD, Harold GT, Kim H, Chamberlain P. Drug Use Trajectories After a Randomized Controlled Trial of MTFC: Associations with Partner Drug Use. J Res Adolesc. 2014 Mar 1;24(1):40-54. doi: 10.1111/jora.12077. PMID 24729667